CLINICAL TRIAL: NCT03972839
Title: Comparison of Two D-Dimers Dosing Techniques : LIATEST DDI PLUS (STAGO) Versus VIDAS D-DIMERS (BIOMERIEUX)
Brief Title: Comparison of Two D-Dimers Dosing Techniques
Acronym: COMPADDI
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0034
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2019-03

CONDITIONS: Blood Coagulation Disorder
Keywords: Blood Coagulation; DDimers
MeSH Terms: conditions — Blood Coagulation Disorders; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- D-Dimers patients: population recruited in Brest for a period of 1 year: patients for whom a dose of VIDAS D-dimers is prescribed (approximately 3700 patients)

SUMMARY:
Study of the possibility of substitution of the automated STAGO D-Dimers method with the semi-automated VIDAS method, which is more expensive, longer to implement and requires the use of a dedicated automaton.

DETAILED DESCRIPTION:
To compare D-Dimer assay techniques in the exclusion of VTE (Thromboembolic Venous Disease):• BIOMERIEUX: D-Dimers VIDAS (considered as reference technique)• STAGO: D-Di PlusOn a population of patients recruited in Brest for a period of 1 year: patients for whom a dosage of VIDAS D-dimers is prescribed (approximately 3700 patients)

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom a dosage of D-Dimers VIDAS is prescribed in the context of a suspicion of VTE at Brest CHRU.
* No opposition formulated.

Exclusion Criteria:

* Curative dose anticoagulant treatment whatever the indication,
* Pregnancy in progress,
* Follow-up at 3 months not possible,
* Patient refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient population recruited in Brest for a period of 1 year: patients for whom a dose of VIDAS D-dimers is prescribed (approximately 3700 patients)
Sampling Method: Non-Probability Sample
Enrollment: 3027 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Biomerieux D-Dimer level | at the inclusion
  quantification of Biomerieux D-Dimer level (VIDAS)
Stago D-Dimer level | at the inclusion
  quantification of Biomerieux D-Dimer level (STAGO)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France